CLINICAL TRIAL: NCT02765230
Title: Interocular Anatomical and Visual Functional Differences in Pediatric Patients With Unilateral Cataracts at 3 Months Post-surgery: A Cross-sectional Study
Brief Title: An Interocular Comparative Study of Unilateral Cataract
Status: Completed | Type: Observational
Sponsor: Sun Yat-sen University (Other)
Collaborators: Ministry of Health, China (Other Government)
Responsible Party: Principal Investigator, Haotian Lin, Principal Investigator, Home for Cataract Children, Zhongshan Ophthalmic Center, Sun Yat-sen University
Other Study IDs: CCPMOH2016-China-3
Record Dates: First submitted 2016-05-03; First posted 2016-05-06 (Estimated); Last update posted 2016-05-06 (Estimated); Status verified 2016-05

CONDITIONS: Cataract
MeSH Terms: conditions — Cataract

STUDY DESIGN:
Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes

SUMMARY:
The purpose of this cross-sectional study is to compare bilateral anterior segment parameters, macular thickness, and BCVA at 3 months after uncomplicated unilateral pediatric cataract extraction with primary IOL implantation to explore any possible interocular differences and their possible relationships.

DETAILED DESCRIPTION:
Great advances have been made in managing pediatric cataracts during the last several decades; these advances have contributed to a decrease in the incidence of postoperative complications and improvement in visual outcomes.Early cataract removal and replacement with an intraocular lens (IOL) represent the most appropriate treatments to avoid irreversible amblyopia.Although screening and timely surgical intervention play a key role in improved best corrected visual acuity (BCVA) among pediatric patients with cataracts, determining the prognosis for an individual remains difficult, particularly for unilateral cataract.

Few studies have focused on the interocular differences in ocular anatomic parameters other than axial length in unilateral pediatric cataract after surgery, the significance of which for the possible interocular visual functional difference remains unclear. Therefore, the investigators conducted this cross-sectional study to compare bilateral anterior segment parameters, macular thickness, and BCVA at 3 months after uncomplicated unilateral pediatric cataract extraction with primary IOL implantation to explore any possible interocular differences and their possible relationships.

ELIGIBILITY:
Inclusion Criteria:

* Children with uncomplicated surgeries
* Children who were younger than 10 years old
* Children with unilateral total cataract

Exclusion Criteria:

* Premature birth
* Microphthalmia
* Micro-or Megalocornea
* Keratoconus
* Glaucoma
* Traumatic or complicated cataracts
* Vitreous and retinal diseases
* Any previous surgeries

Max Age: 10 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: All of the registered children of CCPMOH were diagnosed by anterior segmental photography to confirm the morphology, location, and degree of cataract after pupil dilation. Fifty-three pediatric patients (53 cataract eyes and 53 contralateral normal eyes) with uncomplicated unilateral total cataract were selected 3 months after surgery from the CCPMOH.
Sampling Method: Probability Sample
Enrollment: 53 (Actual)
Dates: Start 2014-01; Primary Completion 2016-01 (Actual); Study Completion 2016-01 (Actual)

PRIMARY OUTCOMES:
Interocular anatomical parameters in pediatric unilateral cataract patients measured by pentacam | Baseline
  The Parameters are measured by pentacam (Oculus Inc., Wetzlar, Germany), a rotating Scheimpflug camera.
Visual function in pediatric unilateral cataract patients measured by Teller Acuity Cards | Baseline
  The visual function is measured by Teller Acuity Cards (Stereo Optical Company, Inc., IL, USA).

CONTACTS AND LOCATIONS:
Overall Officials: Haotian Lin, M.D., Ph.D, Principal Investigator — Zhongshan Ophthalmic Center, Sun Yat-sen University; Yizhi Liu, M.D., Ph.D, Study Chair — Zhongshan Ophthalmic Center, Sun Yat-sen University; Weirong Chen, M.D., Study Director — Zhongshan Ophthalmic Center, Sun Yat-sen University
Locations (1):
- Zhongshan Ophthalmic Center, Sun Yat-sen University, Guangzhou, Guangdong, China

REFERENCES:
- [Background] Hutcheson KA. Application of new ophthalmic technology in the pediatric patient. Curr Opin Ophthalmol. 2007 Sep;18(5):384-91. doi: 10.1097/ICU.0b013e328244e07e. PMID 17700231
- [Background] Lin H, Chen W, Luo L, Congdon N, Zhang X, Zhong X, Liu Z, Chen W, Wu C, Zheng D, Deng D, Ye S, Lin Z, Zou X, Liu Y. Effectiveness of a short message reminder in increasing compliance with pediatric cataract treatment: a randomized trial. Ophthalmology. 2012 Dec;119(12):2463-70. doi: 10.1016/j.ophtha.2012.06.046. Epub 2012 Aug 24. PMID 22921386
- [Derived] Long E, Chen J, Liu Z, Lin Z, Cao Q, Zhang X, Li X, Luo L, Lin H, Chen W, Liu Y. Interocular anatomical and visual functional differences in pediatric patients with unilateral cataracts. BMC Ophthalmol. 2016 Nov 3;16(1):192. doi: 10.1186/s12886-016-0371-5. PMID 27809833
- See also: Description Home page of Zhongshan Ophthalmic Center — http://www.gzzoc.com/